CLINICAL TRIAL: NCT06251479
Title: Study of the Dynamics of Verbal and Non-verbal Interaction in Healthy Subjects, Through the Recording of Body Movements and Non-invasive Neurophysiological Techniques
Acronym: OMNIBUS2023
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Caterina Formica, Caterina Formica, PhD, PSY, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: OMNIBUS2023
Record Dates: First submitted 2023-12-28; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Neuroscience; Neuromodulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A group behavioral 1 (Experimental): The first group will perform perceptual and verbal and non-verbal motor execution tasks, while behavioral measurement techniques will be used.
  Interventions: Behavioral: behavioral 1
- B group behavioral 2 (Experimental): The second group will perform the same tasks as group A and will be subjected to the same measurements as group A. Differently from group A, the members of group B will perform the experimental tasks together with another participant.
  Interventions: Behavioral: behavioral 2
- C group neuromoulation 1 (Experimental): The third group is identical to group A except that neurophysiological measurement techniques will also be applied.
  Interventions: Device: neuromodulation 1
- D group neuromodulation 2 (Experimental): The fourth group is identical to group B except that neurophysiological measurement techniques will also be applied.
  Interventions: Device: neuromodulation 2

INTERVENTIONS:
Behavioral: behavioral 1 — verbal and non verbal tasks
  Arms: A group behavioral 1
Behavioral: behavioral 2 — verbal and non verbal tasks with other partecipants
  Arms: B group behavioral 2
Device: neuromodulation 1 — registration with neurophysiological tecniques during verbal and non verbal tasks
  Arms: C group neuromoulation 1
Device: neuromodulation 2 — registration with neurophysiological tecniques during verbal and non verbal tasks with other partecipants
  Arms: D group neuromodulation 2

SUMMARY:
Based on study literature, the investigators can say that our study aims to give an explanation not only from a behavioral point of view but also with respect to what are the neuronal mechanisms underlying our ability to perceive and analyze our own and others' actions. This is essential to fully understand the complexity of our social behaviors. The knowledge of these mechanisms has a high value and relevant implications for many research fields both within and outside the neurosciences. The project aims to study the neurobehavioral correlates of verbal and non-verbal communication. Through the use of non-invasive behavioral and neurophysiological techniques, the study intends to highlight the neurobehavioral markers that allow to quantify the temporal evolution of communication dynamics in healthy subjects.

DETAILED DESCRIPTION:
Based on study literature, the investigators can say that our study aims to give an explanation not only from a behavioral point of view but also with respect to what are the neuronal mechanisms underlying our ability to perceive and analyze our own and others' actions. This is essential to fully understand the complexity of our social behaviors. The knowledge of these mechanisms has a high value and relevant implications for many research fields both within and outside the neurosciences. The project aims to study the neurobehavioral correlates of verbal and non-verbal communication. Through the use of non-invasive behavioral and neurophysiological techniques, the study intends to highlight the neurobehavioral markers that allow to quantify the temporal evolution of communication dynamics in healthy subjects.

1. the investigators intend to verify whether individual differences in the ability to discriminate the verbal and non-verbal signals of others are reflected in significant differences in the way the same actions are performed.
2. the investigators intend to quantify the behavioral variables during the execution of the action and observe how these are modified in the passage from a single execution to an interaction context.
3. the investigators intend to study how the interactive context influences the cerebral and cortico-muscular oscillatory dynamics during the preparation of the action.
4. the investigators intend to verify whether the activity of the motor system contributes not only to the execution of the action but also, if and, if so, to the perception of the actions of others

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18 and 55 years
* written informed consent
* healthy subjects

Exclusion Criteria:

* epilepsy or at risk of epileptic seizures,
* cardiac pacemaker wearers,
* presence of an implanted infusion pump,
* metal plaques in the skull or metal objects in the eye and skull taking neuroleptic drugs or tricyclic antidepressants,
* migraine or at risk of developing this disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2026-08-16 (Estimated)

PRIMARY OUTCOMES:
Embodiment Scale | 1 hour
  patients have to experience rubber hand illusion first with a silicon and and second with a robotic hand. the embodiment variance is evaluted in the two condition with the embofiment scale

SECONDARY OUTCOMES:
Embodiment Scale | 1 hour
  patients have to experience with a single-pulse Transcranial magnetic stimulation during seeing a visual cue where a human hand is stung. the questionnaire evalute the embodiment variance

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy